CLINICAL TRIAL: NCT01510613
Title: An Open-label, Phase II Study of Pomalidomide and Dexamethasone (PDex) for Previously Treated Patients With AL Amyloidosis.
Brief Title: Pomalidomide and Dexamethasone (PDex) in AL Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giampaolo Merlini, Director, Amyloidosis Research and Treatment Center, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-007-IT; 2011-001787-22 (EudraCT Number)
Record Dates: First submitted 2012-01-11; First posted 2012-01-16 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Primary Amyloidosis of Light Chain Type
Keywords: Pomalidomide; Dexamethasone; treatment; AL amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pomalidomide and Dexamethasone (Experimental)
  Interventions: Drug: Pomalidomide and Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide and Dexamethasone — Pomalidomide: 2-4mg/day, every day in cycles of 28 days until progression or unacceptable toxicity Dexamethasone: 20-40mg/week, on days 1, 8, 15, 22 in cycles of 28 days until progression or unacceptable toxicity

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of Pomalidomide and Dexamethasone in patients who did not achieve a complete response after initial treatment with both an alkylating agent (Melphalan or Cyclophosphamide) and Bortezomib. Patients who received 1 previous treatment without achieving a complete response (CR), but who could not be treated with alkylators and/or Bortezomib due to contraindications, will be included.

DETAILED DESCRIPTION:
This will be a phase II open-label single-arm dose-escalation study. Patients with systemic AL amyloidosis who did not achieve a complete response after initial treatment with both an alkylating agent (Melphalan or Cyclophosphamide) and Bortezomib will be enrolled. Patients who received 1 previous treatment, but who could not be treated with alkylators and/or Bortezomib due to contraindications, will be eligible. Twenty-eight patients will be enrolled in the study. The patients will be treated with the combination of Pomalidomide and Dexamethasone given orally in 28 day cycles continuously, i.e. until hematologic or organ progression or unacceptable toxicity. There will be 2 dose levels of Pomalidomide (2 and 4 mg/day). A standard 3+3 dose escalation design will be used. If less than 2 of 6 patient experience dose limiting toxicity at dose level 1, then all other patients will be treated at dose level 2. There will be 2 dose levels also for Dexamethasone (20 and 40 mg/week). The dose of dexamethasone will be adjusted on an individual basis, considering fluid retention and repetitive ventricular arrhythmias at baseline, as well as Dexamethasone-related adverse events. The study comprises 3 periods: screening, treatment (with evaluations of response at the end of every single cycle) followed by the end-of-treatment evaluation and follow-up. After giving written informed consent, subjects will be evaluated for eligibility for enrollment in the study and baseline evaluations will be performed. Treatment will be continued until progression or unacceptable toxicity is observed. After treatment discontinuation, patients will be followed for survival and any possible Second Primary Malignancies signals for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years.
* Diagnosis of systemic AL amyloidosis.
* Symptomatic organ (heart, kidney, liver, peripheral nervous system, or soft tissue) involvement.
* Patients achieving less than complete response after initial treatment with an alkylating agent (melphalan or cyclophosphamide) and bortezomib. Patients with AL amyloidosis who received 1 previous treatment, but who could not be treated with alkylators and/or bortezomib due to contraindications, will be eligible.
* Measurable disease: difference between amyloidogenic (involved) and uninvolved free light chains (dFLC) > 50 mg/L.
* Hb ≥ 10 g/dL
* ANC ≥ 1500/uL.
* Platelet count ≥ 100000/uL.
* eGFR ≥ 30 mL/min per 1.73 m2.
* Performance status (ECOG) < 3.
* Total bilirubin < 2.5 mg/dL.
* Alkaline phosphatase < 5 × url.
* ALT < 3 × url.
* Female: FCBP must have two negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug. The subject may not receive study drug until the Investigator has verified that the results of these pregnancy tests are negative. Will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure. Must agree to abstain from donating blood during study participation and for at least 28 days after discontinuation from the study.
* Male: Must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy. Will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure. Must agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation from the study.

During study participation and for 28 days following discontinuation from the study:

* All subjects: No more than a 28-day supply of study drug will be dispensed at a time.
* Female: FCBP with regular cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at study discontinuation, and at day 28 following discontinuation from the study. If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study discontinuation, and at days 14 and 28 following discontinuation from the study. In addition to the required pregnancy testing, the Investigator must confirm with FCBP that she is continuing to use two reliable methods of birth control at each visit. Counseling about pregnancy precautions and the potential risks of fetal exposure must be conducted at a minimum of every 28 days. During counseling, subjects must be reminded to not share study drug and to not donate blood. Pregnancy testing and counseling must be performed if a subject misses her period or if her pregnancy test or her menstrual bleeding is abnormal. Study drug treatment must be discontinued during this evaluation. Females must agree to abstain from breastfeeding during study participation and for at least 28 days after discontinuation from the study.
* Male: Counseling about the requirement for latex condom use during sexual contact with females of childbearing potential and the potential risks of fetal exposure must be conducted at a minimum of every 28 days. During counseling, subjects must be reminded to not share study drug and to not donate blood, sperm, or semen.

Exclusion Criteria:

* Amyloid-specific syndrome, such as carpal tunnel syndrome or skin purpura as the only evidence of disease.
* New York Heart association (NYHA) class IV.
* Known positivity for HIV or active hepatitis infection.
* Pregnant or nursing women (men must agree to use an acceptable method for contraception for the duration of the study).
* Uncontrolled infections.
* Other active malignancies.
* Patient has a prior history of thrombosis or venous thromboembolism or pulmonary embolism.
* Known hypersensitivity to thalidomide or lenalidomide including development of erythema.
* Previous or ongoing psychiatric illness (with the exclusion of reactive depression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of PDex | evaluation made at the end of each 28 days cycle
  To evaluate the efficacy of PDex in patients who did not achieve a complete response after initial treatment with both an alkylating agent (Melphalan or Cyclophosphamide) and Bortezomib.

SECONDARY OUTCOMES:
Safety of PDex | evaluation made at the end of each 28 days cycle
  to assess the safety of PDex combination and to assess the survival of AL Amyloidosis patients treated with PDex.

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Merlini, Prof., Principal Investigator — Centro per lo Studio e la Cura delle Amiloidosi Sistemiche - Fondazione IRCCS Policlinico S.Matteo
Locations (1):
- Centro per lo Studio e la Cura delle Amiloidosi Sistemiche - Fondazione IRCCS Policlinico S.Matteo, Pavia, Italy

REFERENCES:
- [Background] Merlini G, Seldin DC, Gertz MA. Amyloidosis: pathogenesis and new therapeutic options. J Clin Oncol. 2011 May 10;29(14):1924-33. doi: 10.1200/JCO.2010.32.2271. Epub 2011 Apr 11. PMID 21483018
- [Background] Palladini G, Russo P, Lavatelli F, Nuvolone M, Albertini R, Bosoni T, Perfetti V, Obici L, Perlini S, Moratti R, Merlini G. Treatment of patients with advanced cardiac AL amyloidosis with oral melphalan, dexamethasone, and thalidomide. Ann Hematol. 2009 Apr;88(4):347-50. doi: 10.1007/s00277-008-0600-y. Epub 2008 Sep 9. PMID 18779964
- [Background] Lacy MQ, Hayman SR, Gertz MA, Dispenzieri A, Buadi F, Kumar S, Greipp PR, Lust JA, Russell SJ, Dingli D, Kyle RA, Fonseca R, Bergsagel PL, Roy V, Mikhael JR, Stewart AK, Laumann K, Allred JB, Mandrekar SJ, Rajkumar SV. Pomalidomide (CC4047) plus low-dose dexamethasone as therapy for relapsed multiple myeloma. J Clin Oncol. 2009 Oct 20;27(30):5008-14. doi: 10.1200/JCO.2009.23.6802. Epub 2009 Aug 31. PMID 19720894
- [Background] Avet-Loiseau H, Soulier J, Fermand JP, Yakoub-Agha I, Attal M, Hulin C, Garderet L, Belhadj K, Dorvaux V, Minvielle S, Moreau P; IFM and MAG groups. Impact of high-risk cytogenetics and prior therapy on outcomes in patients with advanced relapsed or refractory multiple myeloma treated with lenalidomide plus dexamethasone. Leukemia. 2010 Mar;24(3):623-8. doi: 10.1038/leu.2009.273. Epub 2010 Jan 14. PMID 20072152
- [Derived] Palladini G, Milani P, Foli A, Basset M, Russo F, Perlini S, Merlini G. A phase 2 trial of pomalidomide and dexamethasone rescue treatment in patients with AL amyloidosis. Blood. 2017 Apr 13;129(15):2120-2123. doi: 10.1182/blood-2016-12-756528. Epub 2017 Jan 27. PMID 28130212
- See also: Related Info — http://www.amiloidosi.it/